CLINICAL TRIAL: NCT02850640
Title: Cost and Medical Care of Patients With Advanced Serious Illness in Singapore (COMPASS) Study
Acronym: COMPASS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Cancer Centre, Singapore (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Other Study IDs: 2015/2781
Record Dates: First submitted 2016-06-09; First posted 2016-08-01 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Cost and Medical Care of Patients with Advanced Serious Illness in Singapore (COMPASS),is a cohort study which aims to capture health care utilization, cost, and quality of life indicators of patients with advanced cancer and their primary caregivers.

DETAILED DESCRIPTION:
The study will recruit 600 patients with advanced cancer, their primary informal caregivers and their treating physicians. Eligible patients will be recruited from study-sites in Singapore and will be followed until death. Patients and their consenting primary informal caregivers will be interviewed first at baseline and then every 3 months thereafter until the patient's death. A post-death interview with primary informal caregiver will be conducted at 8th week and 6 months after the patient's death. As the majority of the care during last year of life is provided by hospices, the eligible patients will be followed as they receive treatment and care at various hospices. Treating physicians of the patients will be invited to take part in the study. They will be asked to answer a survey conducted only once during the duration of the study.

Data on medical expenditures incurred by a patient from diagnosis of advanced cancer until death will be collected. With patient consent, these data will be extracted every 6 months from the time of patient enrolment from relevant databases, including hospitals and hospices.

ELIGIBILITY:
Inclusion Criteria for patients are:

1. Age ≥ 21 years old
2. Singaporean or Singapore Permanent Resident
3. Diagnosis of advanced/ stage IV solid cancer (for non-breast and non-prostate cancer patients). If it is breast or prostate cancer it should be stage IV with metastases to an organ site.
4. Graded 0-2 on the Eastern Cooperative Oncology Group Performance Status
5. Intact cognition (of patients ≥60 years of age) as determined by the Abbreviated Mental Test. If patient fails the cognitive test, he/she continues to be eligible for the study although self-reported data will no longer be collected. The Legal Representative of the patient will be approached for providing consent on behalf of the patient, to allow access to review of patient's medical and billing records

The exclusion criteria for patients are

1. Patients who are not Singaporeans or Singapore Permanent Residents
2. Patients who are graded 3 (confined to bed more than 50% of waking hours) and 4 (completely disabled) on the Eastern Cooperative Oncology Group Performance Status.
3. Patients who are ≤21 years of age

The inclusion criteria for primary informal caregivers are:

1. Age ≥ 21 years old
2. Main person or one of the main providing care to the patient (e.g. accompanying patient for doctor's visits, helping the patient with day to day activities)
3. Main person or one of the main ensuring provision of care (e.g. supervision of foreign domestic worker so that the patient is looked after)
4. Main person or one of the main involved in making decisions regarding treatment the patient receives
5. Patient they are caring for is enrolled in the study

The exclusion criteria for primary informal caregivers are:

a) Foreign domestic workers/ maids will be excluded from this study

The inclusion criteria for physicians are:

1. Age ≥ 21 years old
2. Patients they are treating are enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV cancer patients, their primary informal caregivers and their treating physicians
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-12; Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in overall quality of life among patients through the last year of life. | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess patient's quality of life through FACT-G
Change in anxiety and depression among patients through the last year of life | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess patients' anxiety and depression through the Hospital Anxiety and Depression Scale (HADS).
Change in pain severity among patients through the last year of life | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess pain reported by patients through visual analog pain scores
Change in activities of daily living among patients through the last year of life | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess limitations in activities of daily living of patients through OARS Multidimensional Functional Assessment Questionnaire
Change in patient's perceived quality of care during the last year of life | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will describe patients' assessment of their own care using a scale used by Ayanian et al (JCO, 2010) that consists of 13 questions.
Total health care expenditure during the last year of life through analysis of medical bills | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will calculate total health care expenditure during the last year of patient's life as the sum total of expenditures incurred at clinics etc.

SECONDARY OUTCOMES:
Change in patient's awareness of prognosis by asking if the patients believe that their current treatment regimen is likely to cure them of cancer | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess knowledge of disease by asking the extent to which advanced cancer patients understand the severity of their condition and if the patients believe that a treatment regimen is available that could cure them
Change in caregiver burden through the last year of life | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess caregiver burden through modified Caregiver Reaction Assessment Scale Instrument
Change in caregiver's levels of emotional distress through the last year of life | From recruitment to death of patient (baseline, 3 month, 6 months, 9 months, 12 months)
  We will assess caregiver's anxiety and depression through the Hospital Anxiety and Depression Scale (HADS).
Caregiver's perception of patient's end-of-life care assessed after patient's death | 8 weeks bereavement
  We will assess caregiver perceived quality of end-of-life care through Caregiver Evaluation of the Quality of End-Of- Life Care( CEQUEL)
Caregivers bereavement adjustment assessed after patient's death | 6 months bereavement
  Post-patient death bereavement adjustment will be assessed through Brief Grief Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD, MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Shafiq M, Malhotra R, Ozdemir S, Teo I, Malhotra C. Trajectories of Health-related quality of life in patients with Advanced Cancer during the Last Year of Life: findings from the COMPASS study. BMC Palliat Care. 2022 Oct 14;21(1):183. doi: 10.1186/s12904-022-01075-3. PMID 36242033
- [Derived] Ozdemir S, Ng S, Chaudhry I, Teo I, Malhotra C, Finkelstein EA; COMPASS Study Group. Caregiver-Reported Roles in Treatment Decision Making in Advanced Cancer and Associated Caregiving Burden and Psychological Distress: A Longitudinal Study. Med Decis Making. 2023 Feb;43(2):191-202. doi: 10.1177/0272989X221125408. Epub 2022 Sep 16. PMID 36113405
- [Derived] Malhotra C, Bundoc F, Chaudhry I, Teo I, Ozdemir S, Finkelstein E; COMPASS study group. A prospective cohort study assessing aggressive interventions at the end-of-life among patients with solid metastatic cancer. BMC Palliat Care. 2022 May 16;21(1):73. doi: 10.1186/s12904-022-00970-z. PMID 35578270
- [Derived] Teo I, Singh R, Malhotra C, Ozdemir S, Dent RA, Kumarakulasinghe NB, Yeo WL, Cheung YB, Malhotra R, Kanesvaran R, Yee ACP, Chan N, Wu HY, Chin SM, Allyn HYM, Yang GM, Neo PSH, Nadkarni NV, Harding R, Finkelstein EA. Cost of Medical Care of Patients with Advanced Serious Illness in Singapore (COMPASS): prospective cohort study protocol. BMC Cancer. 2018 Apr 23;18(1):459. doi: 10.1186/s12885-018-4356-z. PMID 29688843